CLINICAL TRIAL: NCT07186881
Title: Effect of Changes in Diagnostic Protocols for Unexplained Lymphocytic Meningitis and Meningoencephalitis : A Retrospective Single-centre Study
Brief Title: Evolving Diagnostic Approaches to Undocumented Lymphocytic Meningitis and Meningoencephalitis
Acronym: CHAN-MEE
Status: Enrolling by invitation | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, LEFEVRE Benjamin, Doctor (MD PhD), Central Hospital, Nancy, France
Other Study IDs: CHAN-MEE
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Tick Bites; Encephalitis; Meningitis; Viral Encephalitis
Keywords: Tick bite encephalitis; encephalitis; meningitidis; outcomes; diagnosis
MeSH Terms: conditions — Tick Bites; Encephalitis; Meningitis; Encephalitis, Viral; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Period before the change of practice: We are examining a change in clinical practice within our institution. Prior to this change, testing for tick-borne encephalitis (TBE) was not routinely performed in cases of meningitis and meningoencephalitis. Following the implementation of the new protocol, our infectious diseases team now recommends that all clinicians managing patients with compatible clinical presentations conduct TBE serology.
  The patient cohort described here corresponds to the period preceding this change in practice.
- Period after the change of practice: We are examining a change in clinical practice within our institution. Prior to this change, testing for tick-borne encephalitis (TBE) was not routinely performed in cases of meningitis and meningoencephalitis. Following the implementation of the new protocol, our infectious diseases team now recommends that all clinicians managing patients with compatible clinical presentations conduct TBE serology.
  The patient cohort described here corresponds to the period following this change in practice.
  Interventions: Other: Recommendation from the infectious diseases team

INTERVENTIONS:
Other: Recommendation from the infectious diseases team — No commercial product was evaluated in this study. We are assessing the benefits and consequences of a change in clinical practice implemented at the hospital level. At our institution, it is now recommended that TBE serology be performed in all cases of undocumented meningitis or meningoencephalitis.
  The infectious diseases team at our hospital simply advises the clinicians responsible for patient care to perform this test.
  Groups: Period after the change of practice

SUMMARY:
Tick-borne encephalitis (TBE) is a viral infection transmitted by ticks. TBE is the third most common cause of encephalitis in France. Across France, numerous cases of lymphocytic meningitis remain without a definitive diagnosis, notably at the Nancy University Hospital. The objective of this study is to assess the impact of a change in diagnostic practice on the work-up of undocumented lymphocytic meningitis and meningoencephalitis at Nancy University Hospital.

DETAILED DESCRIPTION:
Tick-borne encephalitis (TBE) is a viral infection transmitted by ticks. It is an emerging infectious disease and has been notifiable in France since 2021. TBE is the third most common cause of encephalitis in France, following herpes simplex virus and varicella-zoster virus infections (ENCEIF data).

According to initial data collected by Santé publique France, eastern France is the most affected region, with over half of the reported cases occurring in the Rhône-Alpes and Alsace regions. However, this infection remains relatively unfamiliar to many clinicians and is infrequently investigated during routine diagnostic procedures.

Across France, numerous cases of lymphocytic meningitis remain without a definitive diagnosis, notably at the Nancy University Hospital, where approximately 150 such cases are recorded annually. It is plausible that a proportion of these cases are secondary to TBE infection.

The hypothesis underlying this study is based on these observations. Diagnostic practices at the Nancy University Hospital are currently evolving. The infectious diseases team is actively working to increase clinicians' awareness of TBE, encouraging them to consider this diagnosis when presented with compatible clinical scenarios. Specifically, in cases suggestive of TBE, the infectious diseases team now routinely recommends testing for this pathogen.

This change in practice may lead to an increased rate of documented TBE cases and potentially improve patient management.

The primary objective of this study is to assess the impact of this change in diagnostic practice on the work-up of undocumented lymphocytic meningitis and meningoencephalitis at Nancy University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have received full information regarding the organisation and conduct of the study
* Adults or children
* Hospitalised in a department of Nancy University Hospital with a diagnosis of lymphocytic meningitis or meningoencephalitis
* Cerebrospinal fluid showing more than 5 cells/mm³, with either a negative FilmArray result or no FilmArray performed

Exclusion Criteria:

* Patients diagnosed with non-lymphocytic meningitis or meningoencephalitis
* Patients with documented lymphocytic meningitis or meningoencephalitis of a known cause (excluding TBE) prior to the date the advisory was issued
* Patients who have expressed opposition to the use of their data for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion Criteria:
  * Individuals who have received full information regarding the organisation and conduct of the study
  * Adults or children
  * Hospitalised in a department of Nancy University Hospital with a diagnosis of lymphocytic meningitis or meningoencephalitis
  * Cerebrospinal fluid showing more than 5 cells/mm³, with either a negative FilmArray result or no FilmArray performed
  Exclusion Criteria:
  * Patients diagnosed with non-lymphocytic meningitis or meningoencephalitis
  * Patients with documented lymphocytic meningitis or meningoencephalitis of a known cause (excluding TBE) prior to the date the advisory was issued
  * Patients who have expressed opposition to the use of their data for this study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
TBE diagnosis | This study compares data from the pre-intervention period (2022-2024) with that from the post-intervention period (2024-2026).
  To measure the impact of revised diagnostic procedures on TBE detection among cases of unexplained clear-fluid meningitis and meningoencephalitis at Nancy University Hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nancy, Brabois Hospital, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated and analysed during the current study are not publicly available due to restrictions by the French law, but are available from the last author on reasonable request at the following email address: b.lefevre@chru-nancy.fr.